### STUDY PROTOCOL

Protocol Version: 1.0

Protocol Date: 15 June, 2025

**Ethics Approval:** 

Approved by IREB, University of Lahore Approval No: UOL/IREB/25/09/0030

Approval Date: June 30, 2025

Title: Static versus Dynamic Wrist-Hand Splints for Wrist Spasticity in subacute Stroke

Patients: A Randomized Clinical Trial

### Introduction

Stroke, or cerebrovascular accident, occurs when blood supply to part of the brain is blocked or a cerebral vessel ruptures, resulting in loss of oxygen and essential nutrients. This often leads to paralysis, weakness, impaired coordination and balance, limited mobility, or even death <sup>(1–3)</sup>. Neurological damage disrupts motor control pathways, commonly manifesting as muscle weakness. Following initial injury, the brain undergoes spontaneous recovery through neural plasticity and reorganization <sup>(4–6)</sup>. Stroke is a leading cause of disability globally, with 24.9 million people living with stroke and 11.6 million new cases reported annually in Western Europe <sup>(7,8)</sup>.

Stroke is classified into ischemic ( $\approx$ 80%) and hemorrhagic types <sup>(9)</sup>. Ischemic stroke results from cerebral artery obstruction causing neuronal apoptosis and necrosis in motor regions, while hemorrhagic stroke involves vessel rupture, increased intracranial pressure, and secondary neuronal damage <sup>(7)</sup>. Clinical symptoms include impaired speech, dysphagia, visual and sensory deficits, cognitive impairments, altered muscle tone with spasticity, and inability to walk or grasp objects <sup>(10)</sup>.

Motor dysfunction, low muscle strength, joint stiffness, muscular hypertonia, and muscle contracture are common complications post-stroke <sup>(11–13)</sup>. Post-stroke upper limb spasticity frequently involves involuntary wrist and finger flexor contraction, limiting muscle lengthening and prehensile grasping <sup>(14,15)</sup> (16,17). Approximately 85% of stroke patients experience delayed upper limb recovery, with wrist spasticity affecting 4–46% in chronic stages <sup>(18,19)</sup>.

Rehabilitation through targeted exercises, occupational therapy, and constrained-induced movement therapy improves motor recovery <sup>(20,21)</sup>. Orthotic interventions, including static and dynamic splints, prevent deformities, relieve spasticity, and enhance hand function <sup>(22,23)</sup>. Dynamic splints utilize springs or pulleys to provide gentle, adjustable stretching, and have shown superior efficacy in reducing spasticity when used 6 hours daily <sup>(24,25)</sup>. Despite evidence supporting both types, direct comparisons remain limited <sup>(26,27)</sup>.

## Rationale

This study evaluates the comparative effectiveness of static and dynamic wrist-hand splints in post-stroke rehabilitation, aiming to provide evidence-based guidance for clinicians to optimize treatment strategies and patient outcomes.

### **Materials and Methods**

**Study Design:** A randomized controlled trial (RCT) compared static versus dynamic wrist-hand splints on spasticity, functional hand recovery, and pain in subacute stroke patients.

**Setting:** Markaz Bahali-E-Mazooran Rehabilitation Center, Faisalabad, with trained physiotherapists and occupational therapists supervising interventions.

**Study Duration:** Nine months; each participant underwent a structured 4-week intervention with assessments at baseline and post-intervention.

**Sample Size:** 25 participants initially targeted; after adjustment for dropout, 20 participants (10 per group) completed the study.

**Sampling Technique:** Purposive sampling; participants randomly assigned to groups via computer-generated randomization.

**Inclusion Criteria:** Adults 30–65 years, diagnosed with hemiplegic stroke within last 6 months, moderate to severe wrist spasticity (MAS  $\geq$ 1).

**Exclusion Criteria:** Severe neurological or musculoskeletal disorders, cognitive impairment, contraindications to splint use, or inability to comply with protocols.

**Outcome Measures:** MAS, pain scores, grip strength, functional outcomes, and patient satisfaction at baseline and week 4.

**Statistical Analysis:** Paired t-tests, Wilcoxon signed-rank tests, Mann-Whitney U tests, and repeated-measures ANCOVA used to evaluate changes and compare groups.

# References

- 1. Bhagavatula S, Chang DSH. Comparing the Efficacy of Various Hand Splints in Post Stroke Recovery: A Brief Literature Review. 2021;10(1).
- 2. Chan RKY. SPLINTING FOR PERIPHERAL NERVE INJURY IN UPPER LIMB. Hand Surg. 2002 Dec;07(02):251–9.
- 3. Grefkes C, Fink GR. Recovery from stroke: current concepts and future perspectives. Neurol Res Pract. 2020 Dec;2(1):17.
- 4. Zheng Y, Liu G, Yu L, Wang Y, Fang Y, Shen Y, et al. Effects of a 3D-printed orthosis compared to a low-temperature thermoplastic plate orthosis on wrist flexor spasticity in chronic hemiparetic stroke patients: a randomized controlled trial. Clin Rehabil. 2020 Feb;34(2):194–204.
- 5. Anwer S, Waris A, Gilani SO, Iqbal J, Shaikh N, Pujari AN, et al. Rehabilitation of Upper Limb Motor Impairment in Stroke: A Narrative Review on the Prevalence, Risk Factors, and Economic Statistics of Stroke and State of the Art Therapies. Healthcare. 2022 Jan 19;10(2):190.
- 6. Salaudeen MA, Bello N, Danraka RN, Ammani ML. Understanding the Pathophysiology of Ischemic Stroke: The Basis of Current Therapies and Opportunity for New Ones. Biomolecules. 2024 Mar 4;14(3):305.

- 7. Cantillo-Negrete J, Carino-Escobar RI, Carrillo-Mora P, Rodriguez-Barragan MA, Hernandez-Arenas C, Quinzaños-Fresnedo J, et al. Brain-Computer Interface Coupled to a Robotic Hand Orthosis for Stroke Patients' Neurorehabilitation: A Crossover Feasibility Study. Front Hum Neurosci. 2021 Jun 7;15:656975.
- 8. Wodu CO, Sweeney G, Kerr A. Exploring the reasons behind the low focus on upper limb rehabilitation in the early stages after a stroke: A qualitative study. Journal of Hand Therapy. 2025 Jan;38(1):52–60.
- 9. Boardsworth K, Rashid U, Olsen S, Rodriguez-Ramirez E, Browne W, Alder G, et al. Upper limb robotic rehabilitation following stroke: a systematic review and meta-analysis investigating efficacy and the influence of device features and program parameters. J NeuroEngineering Rehabil. 2025 Jul 16;22(1):164.
- 10. Demeco A, Foresti R, Frizziero A, Daracchi N, Renzi F, Rovellini M, et al. The Upper Limb Orthosis in the Rehabilitation of Stroke Patients: The Role of 3D Printing. Bioengineering. 2023 Nov;10(11):1256.
- 11. Cui Y, Cheng S, Chen X, Xu G, Ma N, Li H, et al. Advances in the clinical application of orthotic devices for stroke and spinal cord injury since 2013. Front Neurol. 2023 Feb 17;14:1108320.
- 12. Song Q, Qin Q, Suen LKP, Liang G, Qin H, Zhang L. Effects of wearable device training on upper limb motor function in patients with stroke: a systematic review and meta-analysis. J Int Med Res. 2024 Oct;52(10):03000605241285858.
- 13. Hirata J, Yoshimura M, Inoue K. The effects of wrist hand orthosis use on upper limb activity and difficulty in activities of daily living: Influence of material and design differences. Journal of Rehabilitation and Assistive Technologies Engineering. 2025 Jul;12:20556683251372060.
- 14. Pritchard K, Edelstein J, Zubrenic E, Tsao L, Pustina K, Berendsen M, et al. Systematic review of orthoses for stroke-induced upper extremity deficits. Topics in Stroke Rehabilitation. 2019 Jul 4;26(5):389–98.
- 15. Ferrari ALM, Medola FO, Sandnes FE. How Do Orthoses Impact Ease of Donning, Handwriting, Typewriting, and Transmission of Manual Torque? A Study of Three Prefabricated Wrist-Hand Orthoses. J Prosthet Orthot. 2021 Jul;33(3):168–74.
- 16. Risangtuni AG, Suprijanto S, Nazaruddin YY, Mahyuddin AI. Dual-mode 3D printed dynamic wrist driven orthosis for hand therapy exercises. Front Mech Eng. 2023 Nov 22;9:1286304.
- 17. Trotobas C. Restoration of grasping functions through assistive orthoses for individuals with arm paralysis [Internet] [phdthesis]. Université de Montpellier; 2023 [cited 2024 Aug 1]. Available from: https://inria.hal.science/tel-04455138
- 18. Thorsen R, Ferrarin M. A Wearable Open-Source Neuroprosthesis/Neuro-Orthosis for Restoring Hand Function. Sensors. 2025 May 23;25(11):3282.
- 19. Umer U, Mian SH, Moiduddin K, Alkhalefah H. Exploring Orthosis Designs for 3D Printing Applying the Finite Element Approach: Study of Different Materials and

- Loading Conditions. Journal of Disability Research [Internet]. 2023 [cited 2025 Oct 28];2(1). Available from: https://scienceopen.com/hosted-document?doi=10.57197/JDR-2023-0011
- 20. Yang YS, Tseng CH, Fang WC, Han IW, Huang SC. Effectiveness of a New 3D-Printed Dynamic Hand–Wrist Splint on Hand Motor Function and Spasticity in Chronic Stroke Patients. JCM. 2021 Sep 30;10(19):4549.
- 21. Mandeljc A, Rajhard A, Munih M, Kamnik R. Robotic Device for Out-of-Clinic Post-Stroke Hand Rehabilitation. Applied Sciences. 2022 Jan 21;12(3):1092.
- 22. Domenighetti S, Ozelie R. Material Matters: A Comparative Analysis of Hand Immobilization Orthoses Using 3D-Printed, Thermoplastic, and Fiberglass Cast. The Open Journal of Occupational Therapy. 2024 Oct 15;12(4):1–12.
- 23. Oud TAM, Lazzari E, Gijsbers HJH, Gobbo M, Nollet F, Brehm MA. Effectiveness of 3D-printed orthoses for traumatic and chronic hand conditions: A scoping review. Lumenta DB, editor. PLoS ONE. 2021 Nov 18;16(11):e0260271.
- 24. Ledoux ED, Barth EJ. Design, modeling, and preliminary evaluation of a 3D-printed wrist—hand grasping orthosis for stroke survivors. Wearable Technol. 2024;5:e12.
- 25. Wong Y, Ada L, Månum G, Langhammer B. Upper limb practice with a dynamic hand orthosis to improve arm and hand function in people after stroke: a feasibility study. Pilot Feasibility Stud. 2023 Jul 27;9(1):132.
- 26. Agnelli Martinez LB, Martinez RA, Agnelli JAM, Elui VMC. Empirical practical evaluation instrument for thermoplastic materials for orthoses. Cad Bras Ter Ocup. 2023;31:e3544.
- 27. Moisan G, Zong-Hao Ma C. Advances in prosthetics and orthotics. BMC Musculoskelet Disord. 2024 Feb 12;25(1):135, s12891-024-07246-y.
- 28. Huber J, Slone S, Bazrgari B. An evaluation of 3D printable elastics for post stroke dynamic hand bracing: a pilot study. Assistive Technology. 2023 Nov 2;35(6):513–22.
- 29. O'Brien L. Adherence to therapeutic splint wear in adults with acute upper limb injuries: a systematic review. Hand Therapy. 2010 Mar;15(1):3–12.
- 30. Tanczak N, Plunkett TK, Lin S, Kuenzler L, Lau M, Kuah WKC, et al. Feasibility of post-stroke hand rehabilitation supported by a soft robotic hand orthosis in-clinic and athome. J NeuroEngineering Rehabil. 2025 Aug 21;22(1):183.